CLINICAL TRIAL: NCT01898962
Title: A Prospective Investigation of Definitive Targeted Therapy for Solid Malignancies With Oligometastases
Brief Title: Definitive Therapy for Oligometastatic Solid Malignancies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rocky Mountain Cancer Centers (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Carter 2005-01; 1073869 (Other: Western IRB)
Record Dates: First submitted 2013-07-08; First posted 2013-07-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Stage IV or Recurrent Carcinoma or Sarcoma
Keywords: Oligometastases; Metastatic cancer; Stereotactic radiosurgery
MeSH Terms: conditions — Recurrence; Sarcoma; Neoplasm Metastasis | interventions — Radiosurgery; Spermine Synthase; Yttrium-90; Microspheres

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Definitive locoregional treatment (Experimental): All sites of active disease should be treated definitively (with one of the interventions listed below). Definitive treatment does not have to be the same for all sites of disease.
  Interventions: Procedure: Complete Surgical Removal; Radiation: Stereotactic Radiosurgery; Radiation: Ablative external beam radiation dose; Procedure: Subtotal surgical removal plus ablative radiation dose; Radiation: Radioembolization

INTERVENTIONS:
Procedure: Complete Surgical Removal
Radiation: Stereotactic Radiosurgery
  Other Names: Stereotactic radiosurgery (SRS) for extracranial metastases are also known as streotactic body radiotherapy (SBRT)
Radiation: Ablative external beam radiation dose
  Other Names: External Beam Radiation Therapy (EBRT) with prescribed doses ≥ 45 Gy (biologic equivalent dose)
Procedure: Subtotal surgical removal plus ablative radiation dose — Residual tumor or close/positive margins should be followed by ablative radiation doses (by either stereotactic radiosurgery or convential EBRT) to constitute definitive locoregional treatment
  Other Names: tumors surgically debulked with residual disease or close/positive margins followed by ablative radiation doses
Radiation: Radioembolization — radioembolization of the liver with Y-90 microspheres or other site-appropriate techniques
  Other Names: Yttrium-90 (Y-90) microspheres; Y-90 radioembolization; SIR-spheres; TheraSphere

SUMMARY:
Patients with metastatic cancer are usually treated with systemic therapy (treating the entire body) with the assumption that any localized treatment of clinically apparent metastases would not impact survival. In the setting of increasingly effective systemic therapy and limited metastatic disease, aggressive treatment to clinically active sites of disease (alone or in addition to systemic therapy) may improve survival.

DETAILED DESCRIPTION:
Up to recently it has been assumed that in the setting of metastatic solid tumors, locoregional control of clinically apparent metastases does not substantially impact survival due to undetectable micrometastic (clinically not visualized) disease that ultimately lead to treatment failure/progression. However, as more advanced systemic therapy continue to improve control of micrometastatic disease, failures at the original sites of disease remain common. Furthermore, some studies have shown locoregional treatment of limited clinical metastases to actually improve survival. Therefore, the investigators hypothesize that aggressive treatment to clinically active sites of disease (alone or in addition to systemic therapy) may improve survival or alter the course of the disease in some patients with limited metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* 4 or less distinct sites of active disease. Locoregional disease counts as one site
* All sites of disease can safely be encompassed by radiation fields to doses ≥ 45 Gy (biologic equivalent dose) and/or removed completely with surgery and/or completely ablated with other appropriate site-specific techniques.
* sufficient blood cell counts and adequate liver function

Exclusion Criteria:

* Hematologic malignancies
* Distinct sites of disease > 4
* Karnofsky Performance Status < 70
* Unexplained weight loss > 10 %
* HIV, chronic viral hepatitis, or any chronically active infection
* Life expectancy < 6 months for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2005-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Survival | 5 years
  Overall and disease-specific survival, to be assessed at 1, 3, and 5 years.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 5 years
  Time to first progression of disease (regardless of location)
Locoregional disease control | 5 years
  Time to first progression within definitively treated areas
Toxicity | 5 years
  Including grade 2+ toxicity attributable to localized study treatment as well as to systemic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Dennise Carter, MD, Principal Investigator — Rocky Mountain Cancer Centers
Locations (4):
- United States (4):
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers - Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers - Thornton, Thornton, Colorado